CLINICAL TRIAL: NCT03639077
Title: Volumetric Changes and Graft Stability in Lateral Window Sinus Augmentation: A Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9302
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Lateral Window Sinus Augmentation
Keywords: Bone graft; Lateral window approach; Sinus augmentation; Volumetric change
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Allograft bone alone (Experimental)
  Interventions: Device: Allograft bone alone
- Allograft and xenograft mixture (Experimental)
  Interventions: Device: Allograft and xenograft mixture

INTERVENTIONS:
Device: Allograft bone alone — The subject will receive an allograft as graft material of choice for sinus augmentation
  Arms: Allograft bone alone
Device: Allograft and xenograft mixture — The subjects will receive a mixture of allograft and anorganic bovine bone xenograft as graft material of choice for sinus augmentation
  Arms: Allograft and xenograft mixture

SUMMARY:
The purpose of this study is to evaluate the stability and volumetric changes of the grafting materials used for lateral window sinus augmentation. In addition, different variables known to affect bone stability and remodeling with regard to the augmentation procedure will be evaluated. Similarly, implant placement will be performed and results will be evaluated after a period of six months.

DETAILED DESCRIPTION:
This will be a prospective clinical study evaluating the stability and volumetric change of two grafting materials used in lateral window sinus augmentation procedure (anorganic bovine bone xenograft alone compared to a mixture of allograft and anorganic bovine bone xenograft). Participants will have the same surgical treatment of the lateral window sinus augmentation procedure. Participants will have a simultaneous implant placement at the time of sinus augmentation procedure or a delayed implant placement based on the stability of the implant evaluation.

Cone beam computed tomography (CBCT) will be used to evaluate the volumetric changes between two groups of graft material in sinus augmentation procedure at three time points: pre-operatively, two weeks post-operation and six months post-operation. Biopsies will be harvested after six months for histological and histomorphometric analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years old
2. In need of sinus augmentation utilizing lateral window sinus technique
3. Presence of bone height of < 8 mm
4. Patient has good oral hygiene (<40% plaque score)
5. Periodontally stable
6. Willingness to fulfill all study requirements

Exclusion Criteria:

1. Currently smoking > 10 cigarettes / day
2. Pregnant, expecting to become pregnant or lactating mothers
3. Uncontrolled Diabetes Mellitus (HbA1c >7)
4. Medical condition that may influence the outcome (Neurologic or psychiatric disorders, systemic infections)
5. Current use of oral bisphosphonates
6. History of IV bisphosphonates use
7. Poor oral hygiene (plaque score >40% based on O'Leary plaque score)
8. Unmanageable Sinus perforations
9. Significant pathology in the region of interest that may compromise the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Graft volumetric stability change | CBCT taken at 2 weeks after the procedure and 6 months after the procedure of sinus augmentation to assess the volumetric changes of the graft material
  CBCT will be the primary tool to evaluate the volumetric stability of the graft material used in the sinus augmentation procedure

SECONDARY OUTCOMES:
Histomorphometric analysis | After 6 months of sinus augmentation procedure when the implant is placed
  Identify histological differences between two groups of graft material in sinus augmentation procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Graduate Periodotics, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided yet if there will be a possibility to publish the study in a journal.